CLINICAL TRIAL: NCT02542852
Title: A Pilot Phase II Study of a Nucleoside Sparing Regimen of Dolutegravir + Atazanavir/r in HIV-1 Infected Patients With Detectable Viremia (DOLATAV Study)
Brief Title: A Study of a Nucleoside Sparing Regimen in HIV-1 Infected Patients With Detectable Viremia
Acronym: Dolatav
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Castagna Antonella (Other)
Collaborators: Bristol-Myers Squibb (Industry); ViiV Healthcare (Industry)
Responsible Party: Sponsor-Investigator, Castagna Antonella, Sub Investigator, IRCCS San Raffaele
Organization: IRCCS San Raffaele (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Dolatav Study
Record Dates: First submitted 2015-08-03; First posted 2015-09-07 (Estimated); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: HIV-1 Infection
Keywords: HIV-1
MeSH Terms: interventions — Atazanavir Sulfate; Ritonavir; dolutegravir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open label single arm (Experimental): Introduction of treatment regimen with atazanavir 300mg qd + ritonavir 100mg qd + dolutegravir 50mg qd
  Interventions: Drug: atazanavir 300 mg + ritonavir 100 mg + dolutegravir 50 mg

INTERVENTIONS:
Drug: atazanavir 300 mg + ritonavir 100 mg + dolutegravir 50 mg — Switch to single arm treatment atazanavir-ritonavir 300-100 mg + dolutegravir 50 mg therapy for 24 weeks
  Other Names: Reyataz 300 mg + norvir 100 mg + tivicay 50 mg

SUMMARY:
Research ipotesis is to assess the efficacy and safety of a nucleos(t)ide sparing regimen of atazanavir/ritonavir 300 mg /100 mg QD + Dolutegravir 50 mg QD for the management of virological failure in HIV-1 infected patients.

The Primary Objective is to explore the 24-week efficacy of a nucleos(t)ide sparing regimen of atazanavir 300 mg QD/ ritonavir 100 mg QD + Dolutegravir 50 mg QD for the management of virologic failure in HIV-1 infected, integrase inhibitor-naïve subjects.

DETAILED DESCRIPTION:
Study design;

• 24-week prospective, single-arm, monocentric, open label, pilot study Participants will be seen at screening, baseline, day 8 and at week 4, 8, 12, 16, 24.

At each visit the following evaluations will be performed:

* clinical assessment.
* routine laboratory tests (hematological tests and clinical chemistry) including hemochromocytometric examination with leukocytic formula, creatinine, creatine kinase, transaminases, phosphorus, calcium, alkaline phosphatase, total and direct bilirubin, gammaGT, uric acid, lactate dehydrogenase, urine analysis, glucose, lipid profile, HIV-RNA and CD4 cell counts.

Additional blood samples will be collected at each visit for storage and further determinations.

During follow-up, at different timepoints, patients will additionally undergo:

* HbA1c and fasting insulin levels and HOMA-IR determination (baseline, week 12, week 24)
* Adherence assessment (questionnaire and/or pills counts) at week 4, 12 and 24.
* ECG (baseline and week 24)

Protocol virologic failure is defined as

* < 1 log10 decrease in plasma HIV-1 RNA by week 12, with subsequent confirmation, unless plasma HIV-RNA < 200 copies/ml OR
* a confirmed rebound in plasma HIV-RNA levels ≥ 50 copies/ml after prior confirmed suppression to < 50 copies/ml OR a confirmed plasma increase in HIV-1 RNA levels > 1log10 copies/ml above the nadir value where nadir is ≥ 50 copies/ml OR
* a plasma HIV-1 RNA level ≥ 50 copies/ml at week 24

Subjects who meet a protocol-defined virologic failure during follow-up will be discontinued from the study.

Patients who suppress HIV-1 RNA < 50 cp/ml before week 24 and have a viral blip ≥ 50 copies/ml at week 24 will undergo a plasma HIV-1 RNA re-test to confirm the virologic failure. At virologic failure subjects will perform genotypic and phenotypic tests and a plasma determination of ATV and DTG Cthrough.

No changes in study treatment are allowed with the exception of ritonavir (RTV) discontinuation in patients with hyperbilirubinemia and/or gastrointestinal adverse events judged as RTV-related by the Investigator. In this case, subjects will remain on study using the regimen ATV 400mg QD + DTG 50mg QD. The discontinuation of RTV will not be considered as treatment failure.

In subjects with plasma HIV-RNA < 50 copies/ml at week 24, the study treatment will be successively provided by Italian National Health system.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with age more than 18 years
* Willing and able to provide informed consent
* Failing a stable (at least 3 months) antiretroviral therapy (HIV-RNA more than 200 copies/ml)
* Any CD4 cell count
* Virus susceptible to atazanavir, defined as a genotypic mutation score inferior to 15 according to the HIV drug resistance database (Stanford University)
* No previous documented virologic failure during an atazanavir-containing regimen
* No previous exposure to integrase inhibitors
* Absolute neutrophil count (ANC) more than 500/mm3
* Haemoglobin more than 8.0 g/dL
* Platelet count more than 60,000/mm3
* e-GFR> 60 ml/min using CKD-EPI equation

Exclusion Criteria:

* Active AIDS-defining condition at Screening
* Serious illness requiring systemic treatment and/or hospitalization
* Current use of immunomodulant or immunosuppressive drugs
* Requirement for any concomitant medications that are prohibited with any study drugs (protocol section 3.6)
* History or presence of hypersensitivity to any of the active substances or to the excipients
* Alanine aminotransferase (ALT) more than 5 times the upper limit of normal (ULN), OR ALT more than 3xULN and bilirubin more than 1.5xULN (with more than 35 percent direct bilirubin)
* Subjects positive for Hepatitis B at screening (HBsAg positive)
* Subjects with anticipated need for Hepatitis C virus (HCV) therapy during the study
* Presence of moderate or severe hepatic impairment (defined as a Class B or C at Child Pugh Classification) or presence of unstable liver disease (as defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, or persistent jaundice) or known biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Pregnancy or pregnancy wish; breastfeeding

Moreover, all clinical conditions reported as an absolute contraindication in the summary of product characteristics of the study drugs, will be considered as exclusion criteria.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-09; Primary Completion 2016-06 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Primary endpoint - The proportion of patients with undetectable HIV RNA viral load ( < 50 copies/ml) at week 24 | 24 weeks
  The proportion of patients with undetectable HIV RNA viral load ( < 50 copies/ml) at week 24.

SECONDARY OUTCOMES:
proportion of patient with undetactable HIV RNA at week 4 (Virologic efficacy) | 4 week
  proportion of patient with undetactable HIV RNA at week 4
Change from baseline CD4 cell counts (Immunological efficacy) | 4,8,12,16,24 weeks
  Change from baseline CD4 cell counts
Time to achieve undetectability (Virologic efficacy) | Day 8, weeks 4,8,12,16,24
  Time to achieve undetectability
Occurrence of genotyping resistance mutations for PI and INSTI in isolates from patients with virological failure. | 24 week
  Occurrence of genotyping resistance mutations for PI and INSTI in isolates from patients with virological failure.
Atazanavir and Dolutegravir Ctrough (PK evaluation) | Day 8, weeks 4,8,12,16,24
  Atazanavir and Dolutegravir Ctrough
Proportion of patients with adverse events (safety and tolerability). | Day 8, weeks 4,8,12,16,24
  Proportion of patients with adverse events (any grade, proportion of patients with more than or equal than grade 2 AE, proportion of patients with side effects leading to discontinuation, reason for treatment discontinuation.
Changes in lipid, clearance creatinine and glycemic profile from baseline (safety and tolerability) | weeks 4,8,12,16,24
  Changes in lipid, clearance creatinine and glycemic profile from baseline
Change in ECG parameters (safety and tolerability) | 24 week
  Change in ECG parameters
Adherence evaluation | 8,12,16,24 weeks
  Adherence changes since first evaluation using questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Adriano Lazzarin, Prof, Principal Investigator — Ospedale San Raffaele
Locations (1):
- Ospedale San Raffaele Scientific Institute, Milan, Italy

REFERENCES:
- [Background] Eron JJ, Clotet B, Durant J, Katlama C, Kumar P, Lazzarin A, Poizot-Martin I, Richmond G, Soriano V, Ait-Khaled M, Fujiwara T, Huang J, Min S, Vavro C, Yeo J; VIKING Study Group. Safety and efficacy of dolutegravir in treatment-experienced subjects with raltegravir-resistant HIV type 1 infection: 24-week results of the VIKING Study. J Infect Dis. 2013 Mar 1;207(5):740-8. doi: 10.1093/infdis/jis750. Epub 2012 Dec 7. PMID 23225901
- [Background] Rathbun RC, Lockhart SM, Miller MM, Liedtke MD. Dolutegravir, a second-generation integrase inhibitor for the treatment of HIV-1 infection. Ann Pharmacother. 2014 Mar;48(3):395-403. doi: 10.1177/1060028013513558. Epub 2013 Nov 19. PMID 24259658
- [Background] Kozal MJ, Lupo S, DeJesus E, Molina JM, McDonald C, Raffi F, Benetucci J, Mancini M, Yang R, Wirtz V, Percival L, Zhang J, Zhu L, Arikan D, Farajallah A, Nguyen BY, Leavitt R, McGrath D, Lataillade M, The Spartan Study Team. A nucleoside- and ritonavir-sparing regimen containing atazanavir plus raltegravir in antiretroviral treatment-naive HIV-infected patients: SPARTAN study results. HIV Clin Trials. 2012 May-Jun;13(3):119-30. doi: 10.1310/hct1303-119. PMID 22592092
- [Background] Song I, Borland J, Chen S, Lou Y, Peppercorn A, Wajima T, Min S, Piscitelli SC. Effect of atazanavir and atazanavir/ritonavir on the pharmacokinetics of the next-generation HIV integrase inhibitor, S/GSK1349572. Br J Clin Pharmacol. 2011 Jul;72(1):103-8. doi: 10.1111/j.1365-2125.2011.03947.x. PMID 21342217
- [Background] Molina JM, Lamarca A, Andrade-Villanueva J, Clotet B, Clumeck N, Liu YP, Zhong L, Margot N, Cheng AK, Chuck SL; Study 145 Team. Efficacy and safety of once daily elvitegravir versus twice daily raltegravir in treatment-experienced patients with HIV-1 receiving a ritonavir-boosted protease inhibitor: randomised, double-blind, phase 3, non-inferiority study. Lancet Infect Dis. 2012 Jan;12(1):27-35. doi: 10.1016/S1473-3099(11)70249-3. Epub 2011 Oct 18. PMID 22015077
- [Background] SECOND-LINE Study Group; Boyd MA, Kumarasamy N, Moore CL, Nwizu C, Losso MH, Mohapi L, Martin A, Kerr S, Sohn AH, Teppler H, Van de Steen O, Molina JM, Emery S, Cooper DA. Ritonavir-boosted lopinavir plus nucleoside or nucleotide reverse transcriptase inhibitors versus ritonavir-boosted lopinavir plus raltegravir for treatment of HIV-1 infection in adults with virological failure of a standard first-line ART regimen (SECOND-LINE): a randomised, open-label, non-inferiority study. Lancet. 2013 Jun 15;381(9883):2091-9. doi: 10.1016/S0140-6736(13)61164-2. PMID 23769235
- [Result] Cahn P, Pozniak AL, Mingrone H, Shuldyakov A, Brites C, Andrade-Villanueva JF, Richmond G, Buendia CB, Fourie J, Ramgopal M, Hagins D, Felizarta F, Madruga J, Reuter T, Newman T, Small CB, Lombaard J, Grinsztejn B, Dorey D, Underwood M, Griffith S, Min S; extended SAILING Study Team. Dolutegravir versus raltegravir in antiretroviral-experienced, integrase-inhibitor-naive adults with HIV: week 48 results from the randomised, double-blind, non-inferiority SAILING study. Lancet. 2013 Aug 24;382(9893):700-8. doi: 10.1016/S0140-6736(13)61221-0. Epub 2013 Jul 3. PMID 23830355
- [Result] Castagna A, Maggiolo F, Penco G, Wright D, Mills A, Grossberg R, Molina JM, Chas J, Durant J, Moreno S, Doroana M, Ait-Khaled M, Huang J, Min S, Song I, Vavro C, Nichols G, Yeo JM; VIKING-3 Study Group. Dolutegravir in antiretroviral-experienced patients with raltegravir- and/or elvitegravir-resistant HIV-1: 24-week results of the phase III VIKING-3 study. J Infect Dis. 2014 Aug 1;210(3):354-62. doi: 10.1093/infdis/jiu051. Epub 2014 Jan 19. PMID 24446523